CLINICAL TRIAL: NCT02635165
Title: Medico-Economic Analysis of Management of Flail Chest Between Medical Treatment and Surgical Treatment With Stracos
Acronym: EMVOLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01844-43
Record Dates: First submitted 2015-11-22; First posted 2015-12-18 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Polytraumatises With Rib Fractures

ARMS (2):
- Surgical treatment with Stracos (Active Comparator): The patient was placed in the lateral decubitus position. The procedure involved a curvilinear thoracic incision overlying the center of the fractured segments. The intercostal muscles were dissected off the rib on its superior aspect away from the fracture site, and the fracture was then reduced. The investigators then chose the most suitable Stracos, which is to be found in two available sizes, 6 or 9 claws, according to the length of the fracture. The clip chosen was molded according to the shape of the corresponding rib and the claws were crimped using special pliers on and around the fractured rib.The investigators treated only one rib out of two with Stracos, and as for displaced or comminuted fractures, the adjacent rib was wrapped using vicryl suture on the osteosynthesis rib.
  Interventions: Device: Thoracic osteosyntheses with Stracos
- Medical treatment (No Intervention)

INTERVENTIONS:
Device: Thoracic osteosyntheses with Stracos
  Arms: Surgical treatment with Stracos

SUMMARY:
Optimize the management of polytraumatises with flail chest: surgical treatment Stracos by decreasing the length of stay and the late complications: pain chronicles, quality of life, respiratory function

ELIGIBILITY:
Inclusion Criteria:

* Patients with flail chest including bifocal fracture of three or more consecutive ribs in at least two places with or without paradoxical movement
* The surgical procedure was performed in the first 48 hours after admission
* pathology with prognosis for survival 6-month-old inferior

Exclusion Criteria:

* Paraplegia or Tetraplegia
* Patients having the necessity of neurosurgical treatment or reanimation of neurosurgical
* Aorta hematoma or rupture
* ß-HCG positive in women
* titanium allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Average cost hospitalization | 4 weeks
  Average cost hospitalization without the intensive care cost.The cost of the hospitalization will be calculated by adding the cost of the surgery and hospital stay- time of the surgery-The number of Stracos used by patient

SECONDARY OUTCOMES:
length of hospital stays of the intensive care department | 4 weeks
  From the first day to the last day in the intensive care department. Care department - monitoring patients with traumatic hemothorax - lung pulmonary infectious associated -
length of hospital stays | 4 weeks
  From the first day to the last day in the hospital
occurence of pulmonary infection | 12 months of follow up
The vital capacity (VC) | visit 3 months, visit 6 months, visit 12 months after the surgery
  Volume measurement (L)
The expiratory reserve volume (ERV) | visit 3 months, visit 6 months, visit 12 months after the surgery
  Volume measurement (L)
The total lung capacity (TLC) | visit 3 months, visit 6 months, visit 12 months after the surgery
  Volume measurement (L)
Residual volume (RV) | visit 3 months, visit 6 months, visit 12 months after the surgery
  Volume measurement (L)
6 min walk test (6MWT) | visit 3 months, visit 6 months, visit 12 months after the surgery
  Distance measurement (M)
Visual analog scorer for pain | at visit 7 days, 28 days, 3 months, 6 months and 12 months
Patient Global Assessment to measure quality of life | at visit 7 days, 28 days, 3 months, 6 months and 12 months
date of return to work | visit 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University of Poitiers, Poitiers, France